CLINICAL TRIAL: NCT06339021
Title: Evaluation of Neointimal Coverage After Guiding De-escalation of Antiplatelet Treatment in Patients With ST-elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention by Optical Coherence Tomography or Angiography of STEMI Patients
Brief Title: OCT or Angiography Guided De-escalation of DAPT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, MD, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAPT-OCT
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Optical Coherence Tomography; Dual Antiplatelet Therapy; Antiplatelet De-escalation; Neointimal Coverage; ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- OCT-guided PCI and DAPT De-escalation (Experimental): OCT-guided PCI follwed by DAPT de-escalation (aspirin and clopidogrel) 30 days after the DES implantation in STEMI patients
  Interventions: Procedure: OCT-guided PCI; Drug: DAPT de-escalation
- OCT-guided PCI and default DAPT regimen (Experimental): OCT-guided PCI follwed by default DAPT regimen (aspirin and ticagrelor) 30 days after the DES implantation in STEMI patients
  Interventions: Procedure: OCT-guided PCI; Drug: default DAPT regimen
- Conventional angiography-based PCI and DAPT De-escalation (Experimental): Conventional angiography-based PCI follwed by DAPT de-escalation (aspirin and clopidogrel) 30 days after the DES implantation in STEMI patients
  Interventions: Procedure: Conventional angiography-based PCI; Drug: DAPT de-escalation
- Conventional angiography-based PCI and default DAPT regimen (Active Comparator): Conventional angiography-based PCI follwed by default DAPT regimen (aspirin and ticagrelor) 30 days after the DES implantation in STEMI patients
  Interventions: Procedure: Conventional angiography-based PCI; Drug: default DAPT regimen

INTERVENTIONS:
Procedure: OCT-guided PCI — OCT-guided PCI based on MLD MAX algorithm
  Arms: OCT-guided PCI and DAPT De-escalation; OCT-guided PCI and default DAPT regimen
Procedure: Conventional angiography-based PCI — Conventional angiography-based PCI
  Arms: Conventional angiography-based PCI and DAPT De-escalation; Conventional angiography-based PCI and default DAPT regimen
Drug: DAPT de-escalation — Aspirin and clopidogrel 30 days after DES implantation
  Arms: Conventional angiography-based PCI and DAPT De-escalation; OCT-guided PCI and DAPT De-escalation
Drug: default DAPT regimen — Aspirin and ticagrelor 30 days after DES implantation
  Arms: Conventional angiography-based PCI and default DAPT regimen; OCT-guided PCI and default DAPT regimen

SUMMARY:
Optical coherence tomography (OCT) offers a high-resolution intravascular imaging modality to accurately assess vessel and lumen geometry and identify the hallmark of a culprit lesion including plaque disruption and thrombus. In addition, the incorporation of the MLD MAX algorithm into daily practice guides an efficient and easily-memorable workflow for optimized OCT-guided percutaneous coronary intervention (PCI) with drug-eluting stents (DES). Regarding the antithrombotic therapy after revascularization, the 2023 ESC guidelines recommend the P2Y12 receptor inhibitor de-escalation (i.e. switching from ticagrelor to clopidogrel) in ACS patients may be considered as an alternative strategy to the default treatment regimen in order to reduce the risk of bleeding events.

Based on the above conclusions, we designed a single-center, prospective, randomized controlled, exploratory study trial to evaluate whether the utility of OCT for guiding PCI with DES followed by antiplatelet de-escalation therapy could further reduce the stent-induced intimal hyperplasia of STEMI patients after stent implantation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ~ 85 years old adult patients;
2. Patients diagnosed with STEMI and undergoing PCI.
3. Patients able and willing to give written informed consent and to comply with the requirements of this study protocol.

Exclusion Criteria:

1. Prior history of intracranial hemorrhage or ischemic stroke during the past 6 months；
2. Allergy to aspirin or clopidogrel or ticagrelor;
3. Occurrence of major adverse cardiovascular event (MACE) within 30 days after undergoing PCI;
4. Platelet count < 50 × 109/L;
5. Major bleeding during the past 12 months;
6. Any form of oral, long-term anticoagulation therapy;
7. Pregnancy or lactation;
8. Suspected aortic dissection;
9. Coronary CT-negative patients;
10. Life expectancy <1 year;
11. Uncontrolled hypertension, systolic blood pressure (SBP) ≥180 mmHg, and/or diastolic blood pressure (DBP) ≥110 mmHg;
12. Comorbid conditions included the presence of any of the following: cardiogenic shock, chronic congestive heart failure with NYHA classes III or IV, left ventricular ejection fraction (LVEF) < 35% at transthoracic echocardiography, hypotension with SBP < 90mmHg and/or DBP < 60mmHg, severe arrhythmia (including high-degree AV block, sick sinus syndrome, sustained ventricular tachycardia), severe pulmonary insufficiency, pulmonary embolism, hepatic insufficiency due to non-cardiac causes (ALT or AST more than three times the upper limit of the institution's normal reference ranges), cirrhosis, severe renal failure (eGFR < 30ml/min/1.73m2);
13. Surgery plan within 30 days;
14. Psychiatric abnormalities or alcohol dependence;
15. Patients who are participating in other clinical trials;
16. Unable to tolerate 1 month of DAPT;
17. Angiographic triple vessel disease coronary disease;
18. Other situations judged by the investigators not to be suitable for the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Neointimal thickness after DES implantation | At 12-month follow up after PCI
  Stent and luminal cross-sectional areas (CSAs) were measured. Neointimal CSA was calculated as stent CSA minus lumen CSA. Neointimal thickness was measured as the distance between endoluminal surface of neointima and strut, which was obtained at 12-month follow-up.

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | During 12-month follow up
  Defined as a composite endpoints of all-cause death, myofarction, stroke and clinically indicated revascularization
BARC types 2-5 bleeding | During 12-month follow up
  Defined as all BARC type 2-5 bleeding events
In-stent thrombosis | During 12-month follow up
  In-stent thrombosis was defined as new ST elevation with anginal symptoms or an equivalent due to thrombotic occlusion of the stent placed at the culprit lesion confirmed by coronary angiography during the index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Principal Investigator — Shenyang Northern Hospital
Locations (1):
- Northern Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali ZA, Karimi Galougahi K, Thomas SV, Abu-Much A, Chau K, Dakroub A, Shlofmitz ES, Jeremias A, West N, Matsumura M, Mintz GS, Maehara A, Shlofmitz RA. Optical Coherence Tomography-Guided Percutaneous Coronary Intervention: Practical Application. Interv Cardiol Clin. 2023 Apr;12(2):215-224. doi: 10.1016/j.iccl.2022.12.003. Epub 2023 Jan 31. PMID 36922062
- [Background] Giugliano RP, Braunwald E. The year in acute coronary syndrome. J Am Coll Cardiol. 2014 Jan 28;63(3):201-14. doi: 10.1016/j.jacc.2013.10.041. Epub 2013 Nov 13. No abstract available. PMID 24239661
- [Background] Bliden KP, Tantry US, Storey RF, Jeong YH, Gesheff M, Wei C, Gurbel PA. The effect of ticagrelor versus clopidogrel on high on-treatment platelet reactivity: combined analysis of the ONSET/OFFSET and RESPOND studies. Am Heart J. 2011 Jul;162(1):160-5. doi: 10.1016/j.ahj.2010.11.025. Epub 2011 Jun 12. PMID 21742103
- [Background] Capodanno D, Alfonso F, Levine GN, Valgimigli M, Angiolillo DJ. ACC/AHA Versus ESC Guidelines on Dual Antiplatelet Therapy: JACC Guideline Comparison. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2915-2931. doi: 10.1016/j.jacc.2018.09.057. PMID 30522654
- [Background] Cuisset T, Deharo P, Quilici J, Johnson TW, Deffarges S, Bassez C, Bonnet G, Fourcade L, Mouret JP, Lambert M, Verdier V, Morange PE, Alessi MC, Bonnet JL. Benefit of switching dual antiplatelet therapy after acute coronary syndrome: the TOPIC (timing of platelet inhibition after acute coronary syndrome) randomized study. Eur Heart J. 2017 Nov 1;38(41):3070-3078. doi: 10.1093/eurheartj/ehx175. PMID 28510646
- [Background] Sibbing D, Aradi D, Jacobshagen C, Gross L, Trenk D, Geisler T, Orban M, Hadamitzky M, Merkely B, Kiss RG, Komocsi A, Dezsi CA, Holdt L, Felix SB, Parma R, Klopotowski M, Schwinger RHG, Rieber J, Huber K, Neumann FJ, Koltowski L, Mehilli J, Huczek Z, Massberg S; TROPICAL-ACS Investigators. Guided de-escalation of antiplatelet treatment in patients with acute coronary syndrome undergoing percutaneous coronary intervention (TROPICAL-ACS): a randomised, open-label, multicentre trial. Lancet. 2017 Oct 14;390(10104):1747-1757. doi: 10.1016/S0140-6736(17)32155-4. Epub 2017 Aug 28. PMID 28855078
- [Background] Bonello L, Laine M, Kipson N, Mancini J, Helal O, Fromonot J, Gariboldi V, Condo J, Thuny F, Frere C, Camoin-Jau L, Paganelli F, Dignat-George F, Guieu R. Ticagrelor increases adenosine plasma concentration in patients with an acute coronary syndrome. J Am Coll Cardiol. 2014 Mar 11;63(9):872-7. doi: 10.1016/j.jacc.2013.09.067. Epub 2013 Nov 27. PMID 24291273
- [Background] Kim CJ, Park MW, Kim MC, Choo EH, Hwang BH, Lee KY, Choi YS, Kim HY, Yoo KD, Jeon DS, Shin ES, Jeong YH, Seung KB, Jeong MH, Yim HW, Ahn Y, Chang K; TALOS-AMI investigators. Unguided de-escalation from ticagrelor to clopidogrel in stabilised patients with acute myocardial infarction undergoing percutaneous coronary intervention (TALOS-AMI): an investigator-initiated, open-label, multicentre, non-inferiority, randomised trial. Lancet. 2021 Oct 9;398(10308):1305-1316. doi: 10.1016/S0140-6736(21)01445-8. PMID 34627490
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654